CLINICAL TRIAL: NCT01831999
Title: Clinical Monitoring to Facilitate Continuous Care for Substance Abusing Clients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Treatment Research Institute (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Sponsor
Organization: Public Health Management Corporation (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1R01DA030480-01A1 (NIH); 1R01DA030480-01A1 (NIH)
Record Dates: First submitted 2013-03-29; First posted 2013-04-15 (Estimated); Last update posted 2023-03-28 (Actual); Status verified 2023-03

CONDITIONS: Substance-Related Disorders; Mental Disorders
Keywords: Web-based; HIV Assessment; Outreach; Retention; Substance Abuse Treatment
MeSH Terms: conditions — Substance-Related Disorders; Mental Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- RecoveryTrack - Extended Care (RT-E) (Experimental): Counselors will conduct monitoring and feedback sessions using the RecoveryTrack-Extended Care (RT-E) web-based monitoring system for clients newly admitted to Intensive Outpatient (IOP) treatment. Counselors will be instructed to document their reminders, contact attempts, and scheduling of RT-E appointments within a Contact Log incorporated into RT-E. All RT-E sessions will be audio recorded.
  Interventions: Behavioral: RecoveryTrack - Extended Care (RT-E)
- Treatment as Usual (TAU) (No Intervention): Counselors will conduct standard treatment during IOP/OP in this condition. Exceptions to this condition are that counselors will: audio record their first 3 biweekly and subsequent 7 monthly individual in-person sessions; document on a Contact Log outreach attempts; and complete a Counselor Activity Log for client participants. There are several steps that counselors typically take when a client misses a session. Clients are called to reschedule for the same week, if the client doesn't return for their next scheduled session, the counselor sends a letter asking the client to return, etc.

INTERVENTIONS:
Behavioral: RecoveryTrack - Extended Care (RT-E) — Counselors in this condition will be trained on the RecoveryTrack-Extended Care (RT-E) web-based monitoring system so that they are able to navigate the computer application, and implement the clinical content and procedures of the intervention. Counselors will conduct monitoring and feedback sessions using RT-E for clients newly admitted to IOP over a course of eight months. If the client is not attending treatment, counselors will attempt contact over the phone and via other methods. When contacted, the counselor will conduct the RT-E assessment and, as the situation warrants, provide support to reengage the client in treatment or support recovery in other ways mentioned. HIV risk will be assessed as well, with encouragement of testing and referral to HIV specialists as needed.
  Arms: RecoveryTrack - Extended Care (RT-E)

SUMMARY:
Building on the recent advances in telephone supported care, clinical monitoring, and outreach work, the specific aims of the study are to:

1. Develop RecoveryTrack™- ExtendedCare (RT-E), a modified/new version of RecoveryTrack™. The investigators will adapt and finalize the original Web-based RT system, manual, and training to accommodate use by counselors for clients who are no longer attending Outpatient (OP) treatment.
2. Conduct a pilot study to determine the preliminary efficacy of RT-E compared to treatment as usual (TAU) for clients entering Intensive Outpatient (IOP) substance abuse treatment (SAT). In this randomized clinical trial, it is hypothesized that RT-E will positively impact treatment attendance and substance use outcomes. In exploratory analyses, the investigators will also evaluate the comparative impact of RT-E versus TAU on HIV related client behaviors.
3. Evaluate feasibility and counselor and client acceptability of RT-E.
4. Conduct preliminary cost and cost effectiveness analyses comparing RT-E to TAU.

Hypothesis 1: RT-E clients will attend more days of OP treatment than TAU clients. The investigators will compare the two groups on monthly treatment attendance for months 1 through 9. We expect a main effect of group with RT-E clients displaying more attendance than TAU clients.

Hypothesis 2: RT-E clients will have higher rates of abstinence than TAU clients. The investigators will compare abstinence rates at months 3, 6, and 9. Abstinence is a binary variable based on both biological test results and self-reported substance use from the Addiction Severity Index, Version 6 (ASI6). We expect a main effect of group with RT-E clients displaying higher rates of abstinence than TAU clients.

Secondary Analyses:

HIV Risk Scores: The investigators will compare the two groups' Risk Assessment Battery (RAB) HIV risk scores (i.e., total, sex, drug) at month 9.

Use of HIV specialist services: Client attendance charts will be reviewed to compare the two groups on the number of times clients met with a program HIV Specialist at month 9.

Multidimensional Outcomes: The investigators will compare RT-E and TAU clients on multidimensional outcomes using ASI6 summary scores at months 3, 6, and 9.

DETAILED DESCRIPTION:
The goal of the RecoveryTrack Extended Care (RT-E) study is to improve attendance and extended care treatment during outpatient substance abuse treatment (SAT). One way we hope to promote and improve retention in outpatient treatment is to allow the primary counselor to systematically monitor client progress and respond accordingly to enhance the client's progress in outpatient treatment. We have developed an intervention using RecoveryTrack software that allows the counselor to monitor the client while s/he is regularly attending and to helps to guide their treatment; as well as reaching out and monitoring the client when s/he has missed sessions or appears to have dropped out in order to support re-engagement in treatment or recovery in other ways. SAT can serve as a gateway to and provide services for HIV/STI prevention and treatment as well. Thus, monitoring and responding to HIV/STI risk behavior and treatment compliance throughout SAT, and increasing attendance in SAT itself, has the potential for additional personal and public health impact.

Counselors are trained on the RT-E computer application, and learn to implement the clinical content and procedures of the RT-E intervention. Clients then are asked to use the software with participants twice within the first month, and once monthly for 8 months. If clients drop out of treatment or do not show for an appointment, counselors are asked to do "outreach" with the clients to promote re-entry into treatment. We also ask the counselors to keep track of any time that they spend on the project and how much of their own resources to perform outreach. We ask that all sessions be audio recorded and will be rated at a later time. The TAU counselors also audio record their sessions and document their time on a log any outreach attempts. The counselors are asked to perform their usual outreach attempts if a client drops from treatment, and to complete individual sessions without the RT-E computer application.

In total, 25 counselor-participants will be enrolled in RT-E study. All counselors receive incentives throughout participation in the study. The incentives are greater in the RT-E condition reflecting a greater workload than in TAU with payments at the beginning, middle, and end of research participation. The compensation for counselor participants in each condition is as follows: RT-E training takes approximately 4-5 hours over a period of several weeks at the beginning of the study. RT-E counselors are paid $125 upon completing the entire training sequence. RT-E counselors receive supervision by TRI staff in 30 minute sessions about once a month during the 1st 6 months of the study and quarterly thereafter, for a total of approximately 11 sessions. RT-E counselors are paid $15 for each supervision session attended [maximum total = $165].Two times, midway and near the end of the study, RT-E counselors complete the Counselor Acceptability Survey and are reimbursed $20 each time. Each week RT-E counselors completes the Counselor Activity Log and is paid $2 for each one completed during the course of the study [a maximum of $200 for approximately 104 weeks ].RT-E Counselors are paid $30 for each completed and audio-recorded phone outreach session ($25 if completed but not recorded). Total counselor payment for these activities will vary based on number of client participants seen as well as client non-attendance and need for and responsiveness to outreach contact. Two times, midway and near the end of the study, TAU counselors complete the Counselor Acceptability Survey and are reimbursed $20 each time.

In total, 150 client-participants will be enrolled in the RT-E study. These participants will complete a baseline research interview and follow-up interviews 3, 6 and 9 months later, as well as provide urine samples for drug screening (UDSs) at each of the research assessments. Clients will be contacted at the midpoint of each follow-up interval to remind them of the upcoming follow-up appointment and obtain updated locator information. Clients are paid $30 for completing the baseline ASI6, urine drug screen (UDS), and Risk Assessment Battery (RAB); $35 for the 3-month follow-up ASI6, UDS, and Client Acceptability Interview; $40 for the 6-month ASI6 & UDS, and $50 for completing the 9-month ASI6, UDS, RAB, & Client Acceptability Survey. At months 2, 5, and 8, participants receive reminder letters or phone calls about their upcoming follow-up and can earn $5 each of those months by calling TRI and updating their Research Locator Form. All payments are be in cash, unless a check or money order is more practical (e.g., if payment needs to be mailed). Clients are randomly assigned to groups based on their primary counselors' assignment to condition in the study.

ELIGIBILITY:
Inclusion Criteria:

* Client enrolled in outpatient treatment at participating facility and assigned to participating counselor.
* Counselor employed at participating facility.

Exclusion Criteria:

* Client unable to speak English.
* Client too cognitively impaired to give informed consent.
* Clients who do not wish to be audio-recorded during individual sessions.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 139 (Actual)
Dates: Start 2012-06; Primary Completion 2016-02 (Actual); Study Completion 2016-05 (Actual)

PRIMARY OUTCOMES:
Length of Stay | 9 months post-consent
  Client admission and discharge dates will be obtained from the treatment program clinical record and used to calculate length of stay.

SECONDARY OUTCOMES:
HIV Risk Scores | 9 months post-consent
  The investigators will compare the two groups' Risk Assessment Battery (RAB) HIV risk scores (i.e., total, sex, drug) at month 9.
Multidimensional Outcomes | 3, 6, and 9 months post-consent
  We will compare RT-E and TAU clients on multidimensional outcomes using ASI6 summary scores at months 3, 6, and 9.
Rates of Abstinence | Months 3, 6, and 9 post-consent
  Abstinence is a binary variable based on both biological test results and self-reported substance use from the ASI6.
Use of HIV specialist services | 9 months post-consent
  Client attendance charts will be reviewed to compare the two groups on the number of times clients met with a program HIV Specialist at month 9.

CONTACTS AND LOCATIONS:
Overall Officials: John S. Cacciola, Ph.D., Principal Investigator — Treatment Research Institute
Locations (4):
- United States (4):
  - Genesis Counseling Centers, Inc., Collingswood, New Jersey
  - Genesis Counseling Centers, Inc., Marlton, New Jersey
  - New Journeys In Recovery, Philadelphia, Pennsylvania
  - Thomas Jefferson University IOP, Philadelphia, Pennsylvania

IPD SHARING:
Plan to Share IPD: Undecided